CLINICAL TRIAL: NCT00024817
Title: Energy Expenditure, Diet and Body Fat in Children
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 986; R01HL065053 (NIH)
Record Dates: First submitted 2001-09-28; First posted 2001-09-28 (Estimated); Last update posted 2016-07-15 (Estimated); Status verified 2004-08

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Obesity
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Obesity

SUMMARY:
To characterize the pattern of change over a two year period in energy expenditure and energy intake in two cohorts of American Indian (AI) children.

DETAILED DESCRIPTION:
BACKGROUND:

Obesity is highly prevalent in American Indian children, increasing their risk for the development of cardiovascular disease, hypertension and diabetes. Although increasing energy expenditure, through increasing physical activity, and decreasing dietary fat intake should slow the rate of body fat gain, it appears that children actually decrease their physical activity as they mature from pre-to post-pubescence. Several studies have shown that the decline in activity is greater in females than in males, and greater in non-whites than in whites; however, other studies have not supported these findings. Further, there were no data available in American Indian children, which is a population at greatest risk. Additionally, inconsistencies have been reported with respect to the relationship between body weight or body fat and energy intake or dietary fat intake. At the heart of the problem is the difficulty in measuring self-reported physical activity and dietary intake accurately. Accurate self- report measures are necessary for use in the large scale studies that are required to investigate relationships between physical activity and dietary intake and disease. The Healthy People 2000: National Health Promotion and Disease Prevention Objectives include seven objectives emphasizing increasing physical activity in children and adolescents.

DESIGN NARRATIVE:

This study had a combined longitudinal and cross-sectional design in which the investigators modified the best existing methods for the self-report of physical activity and dietary intake in children and adolescents, and evaluated their validity using total energy expenditure (TEE) measured by doubly labeled water (DLW) as the criterion. They then used these methods to measure physical activity and dietary intake in two age cohorts of male and female American Indian children (8-10-years and 11-13-years) at baseline and two years later, with two sets of interim measurements. Change in TEE from baseline to the two-year follow-up was also measured using DLW and the TriTrac accelerometer. Equations for the estimation of percent body fat were cross-validated for this population. The study filled an existing gap by improving existing instruments for the measurement of physical activity and dietary intake in children and adolescents, and provided longitudinal data on change in these variables in the same children over time, plus provided cross-sectional data for each age and gender group to compare to the existing literature.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Ages: 8 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Dates: Start 1999-09; Study Completion 2002-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judith Weber — Arkansas Children's Hospital Research Institute